CLINICAL TRIAL: NCT04397185
Title: Randomized Prospective Trial of Breast Cancer Locator Guided vs. Wire Localized Partial Mastectomy for Breast Cancer
Brief Title: Breast Cancer Locator Guided vs. Wire Localized Partial Mastectomy for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CairnSurgical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BCL IDE
Record Dates: First submitted 2020-05-15; First posted 2020-05-21 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer Female
MeSH Terms: interventions — Mastectomy, Segmental

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Pathologist will be blinded to the study assignment (BCL vs. WL)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Breast Cancer Locator (BCL) (Experimental): Subject randomized to BCL surgical guidance to perform partial mastectomy
  Interventions: Device: Breast Cancer Locator (BCL) guided partial mastectomy
- Wire Localization (WL) (Active Comparator): Subject randomized to WL surgical guidance to perform partial mastectomy
  Interventions: Device: Wire Localized (WL) partial mastectomy

INTERVENTIONS:
Device: Breast Cancer Locator (BCL) guided partial mastectomy — The BCL is a patient-specific, plastic, bra-like form which is placed on the breast to localize the tumor during surgery.
  Arms: Breast Cancer Locator (BCL)
Device: Wire Localized (WL) partial mastectomy — Standard of care procedure
  Arms: Wire Localization (WL)

SUMMARY:
This prospective, multicenter, 1:1 randomized, controlled trial is designed to evaluate the safety and effectiveness of the Breast Cancer Locator (BCL) in subjects with non-palpable invasive breast cancer or ductal carcinoma in situ (DCIS). Subjects will be randomized to breast conserving surgery (BCS) utilizing either the BCL or wire localization (WL) to guide surgery.

DETAILED DESCRIPTION:
The BCL System is intended to be used to guide a surgeon when performing partial mastectomy for breast cancer and to minimize positive margins. The purpose of this study is to provide evidence that the BCL is safe, effective, and non-inferior to the standard of care (WL) in the removal of non-palpable invasive breast cancer and DCIS.

Investigators in the intervention group will be provided with a three dimensional (3D) image of the cancer in the breast which allows them to visualize the closest distance from the tumor to the skin and the chest wall and quantifies those distances. Investigators will also use a BCL, which is a patient specific, plastic, bra-like form that is transiently placed on the breast prior to surgery and allows the Investigator to mark the projected edges of the tumor on the breast skin and to place bracketing wires inside the breast which define the center of the cancer and distances 1 cm from the tumor edges defined by pre-operative supine MRI.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Age > 18 years
* Histologic diagnosis of invasive breast cancer or DCIS
* The surgeon determines that pre-operative tumor localization is required because the tumor cannot be definitively detected by palpation
* The tumor is unifocal or multifocal with satellite lesions < or = 2 cm from primary tumor
* The tumor enhances on prone breast MRI imaging
* The tumor is ≥ 1 cm in diameter on prone breast MRI
* Subject and surgeon agree to perform BCS
* Subject voluntarily provides informed consent

Exclusion Criteria:

* Absolute contraindication to MRI, including presence of implanted electrical device (e.g., pacemaker or neurostimulator), aneurysm clip, or metallic foreign body in or near eyes
* Severe claustrophobia that precludes prone or supine MRI
* Contraindication to use of gadolinium-based intravenous contrast, including life- threatening allergy
* Compromised renal function including chronic, severe kidney disease (GFR < 30 ml/min/1.73m2), or acute kidney injury
* Pregnancy - In women of childbearing potential, a urine pregnancy test will be performed
* Subjects who have received or plan to receive neoadjuvant chemotherapy
* Sternal notch to nipple distance of > 32 cm as measured in a sitting or standing position
* Measurement of widest circumference around breasts and arms > 135 cm for sites using 60cm bore scanners, and measurement of widest circumference around breasts and arms >145 cm for sites using 70 cm bore scanners
* Subjects with known allergy to materials present in the device
* Use of localization with devices other than a localization wire, including intraoperative ultrasound guidance, radiofrequency emitting implants, magnetic seeds, radioactive seeds, and tissue inspection devices (MarginProbe)
* Subject would require > 2 localization wires, if randomized to standard of care
* Subjects with multicentric tumors (additional tumors > 2 cm from primary)
* Subject would require chest wall muscle nerve block as part of the operation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
Positive margin rate | At completion of study recruitment, approximately 18 months after first subject enrolled
  To provide evidence that the positive margin rate following BCS using the BCL is not inferior to the standard of care (WL) for surgical guidance

SECONDARY OUTCOMES:
Specimen volumes | At completion of study recruitment, approximately 18 months after first subject enrolled
  To compare specimen volumes for women randomized to BCL vs. WL-guided BCS
Re-excision rate | At completion of study recruitment, approximately 18 months after first subject enrolled
  To compare re-excision rate for women randomized to BCL vs. WL-guided BCS
Cancer localization rate | At completion of study recruitment, approximately 18 months after first subject enrolled
  To compare cancer localization rate for women randomized to BCL vs. WL-guided BCS
Operative times | At completion of study recruitment, approximately 18 months after first subject enrolled
  To compare operative times for women randomized to BCL vs. WL-guided BCS
Adverse event rate | At completion of study recruitment, approximately 18 months after first subject enrolled
  To compare adverse event rate for women randomized to BCL vs. WL-guided BCS
Rate of additional shave biopsies | At completion of study recruitment, approximately 18 months after first subject enrolled
  To compare rate of additional shave biopsies for women randomized to BCL vs. WL-guided BCS
Costs of care | At completion of study recruitment, approximately 18 months after first subject enrolled
  To compare costs of care for women randomized to BCL vs. WL-guided BCS

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Gass, MD, Principal Investigator — Women & Infants Hospital
Locations (23):
- United States (19):
  - Arizona Center for Cancer Care, Scottsdale, Arizona
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Tufts Medical Center, Boston, Massachusetts
  - Mass General/North Shore Center for Outpatient Care, Danvers, Massachusetts
  - Steward Medical Group, Easton, Massachusetts
  - Hennepin Healthcare, Minneapolis, Minnesota
  - Cheshire Medical Center, Keene, New Hampshire
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Catholic Medical Center, Manchester, New Hampshire
  - St. Joseph Hospital, Nashua, New Hampshire
  - Summit Health, Florham Park, New Jersey
  - St. Peter's Hospital, Albany, New York
  - Columbia University Irving Medical Center and New York-Presbyterian Hospital, New York, New York
  - Women and Infants Hospital, Providence, Rhode Island
  - Kent Hospital, Warwick, Rhode Island
  - MD Anderson Cancer Center, Houston, Texas
  - Rutland Regional Medical Center, Rutland, Vermont
  - Inova Schar Cancer Institute, Fairfax, Virginia
- LKH Feldkirch, Feldkirch, Austria
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- United Kingdom (2):
  - Basildon University Hospital, Basildon
  - Manchester University NHS, Manchester